CLINICAL TRIAL: NCT01363089
Title: Open Label, 2-Way Crossover Study to Assess the PK of Intranasal Ketorolac Tromethamine and to Assess the Effects of a Single Dose of Oxymetazoline Hydrochloride on the PK of Intranasal Ketorolac Tromethamine in Healthy Male Subjects
Brief Title: Study to Assess the PK of Ketorolac Tromethamine Intranasal and to Assess the Effects of a Oxymetazoline Hydrochloride on the PK of Ketorolac Tromethamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROX 2006-03
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Assess Pharmacokinetics of Ketorolac Tromethamine Intranasal and Assess Effects of a Oxymetazoline Hydrochloride on the PK of Ketorolac Tromethamine
MeSH Terms: interventions — Ketorolac Tromethamine; Oxymetazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketorolac tromethamine (Experimental)
  Interventions: Drug: Ketorolac tromethamine
- Oxymetazoline hydrochloride (Experimental)
  Interventions: Drug: Oxymetazoline hydrochloride

INTERVENTIONS:
Drug: Ketorolac tromethamine — 30 mg of intranasal ketorolac tromethamine (one 100 µL spray into each nostril of a 15%, pH 7.2 solution)
  Arms: Ketorolac tromethamine
Drug: Oxymetazoline hydrochloride — Single intranasal dose of oxymetazoline hydrochloride (Afrazine®) (3 sprays of a 0.05% solution into each nostril) followed 30 minutes later by 30 mg of intranasal ketorolac tromethamine (one 100 µL spray into each nostril of a 15%, pH 7.2 solution)
  Arms: Oxymetazoline hydrochloride

SUMMARY:
This was an open label, two way crossover study in healthy male subjects. Two treatments were administered to each subject, one treatment per study period, in a randomized manner. Subjects remained resident in the Clinical Unit from the evening of Day 1 until the morning of Day 2 of each period and there was a washout period of at least 2 days between treatments. A post study medical examination was performed prior to discharge in Period 2.

The objective of this study was to assess the effects of a single dose of intranasal oxymetazoline hydrochloride on the pharmacokinetics of intranasal ketorolac in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject was male and aged 18 to 62 years inclusive
* Male subjects with female partners of child bearing potential must have consented to use a medically acceptable method of contraception (oral or implanted contraceptive hormones, intrauterine device or surgical sterilization plus condom or diaphragm with spermicidal agent) throughout the study period
* Subject had given signed informed consent
* Subject was within 20% of normal weight for his height and body build according to the table of "Desirable Weights for Men and Women" (Metropolitan Life Insurance Co. 1999)
* Subject's medical history was considered normal, with no clinically significant abnormalities
* Subject was considered to be in good health in the opinion of the Investigator, as determined by a pre-study physical examination with no clinically significant abnormalities, vital signs within normal ranges and an electrocardiogram (ECG) with no clinically significant abnormalities
* Subject's pre-study clinical laboratory findings were within normal range or if outside of the normal range were not deemed clinically significant in the opinion of the Investigator
* Subject had bilateral patent nasal airways at screening and Day 1 as assessed by the Investigator
* Subject had a body weight of at least 60 kg

Exclusion Criteria:

* Subject had had a clinically significant illness in the 4 weeks before screening
* Subject used prescribed medications in the 3 weeks prior to dosing or over the counter preparations for 7 days prior to dosing, except paracetamol which was allowed up to 48 hours (h) prior to dosing. Use of multivitamins was permitted
* Subject had a significant history of drug/solvent abuse, or a positive drugs of abuse test at screening
* Subject had a history of alcohol abuse or currently drank in excess of 28 units per week
* Subject currently used tobacco or had a history of smoking within the past 5 years
* Subject was in the opinion of the Investigator not suitable to participate in the study
* Subject had participated in any clinical study with an investigational drug/device within 3 months prior to dosing
* Subject had a positive human immunodeficiency virus (HIV), hepatitis B or hepatitis C screen
* Subject had had a serious adverse reaction or significant hypersensitivity to any drug
* Subject had donated 500 mL or more of blood within the 3 months prior to screening
* Subject had any history of co-existing nasal polyps, NSAID sensitivity and asthma
* Subject had an allergic reaction to aspirin or other NSAIDs
* Subject currently had an upper respiratory tract infection or other respiratory tract condition that could interfere with the absorption of the nasal spray or with the assessment of AEs
* Subject had any suspicion of rhinitis medicamentosa (chronic daily use of topical decongestants)
* Subject had used a monoamine oxidase inhibitor in the 14 days prior to study entry
* Subject had an active peptic ulcer disease, gastrointestinal bleeding or perforation, or a history of peptic ulcer disease or gastrointestinal bleeding
* Subject had anemia due to unexplained or known gastrointestinal bleeding
* Subject had a history of asthma or any other chronic pulmonary disorder
* Subject had renal impairment or a risk of renal failure due to volume depletion
* Subject had a previous history of nasal surgery

Ages: 18 Years to 62 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Cmax (the maximum observed plasma concentration) | All PK parameters were assessed using blood samples collected pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, and 24 hours post-dose
  Pharmacokinetic analysis by standard model independent methods was performed by a pharmacokineticist using WinNonlin Professional. Actual blood sampling times for ketorolac assay were converted to a time from dosing (elapsed time). Elapsed times were listed by subject for each treatment, together with the individual plasma concentrations of ketorolac.
Tmax (the time to maximum concentration) | All PK parameters were assessed using blood samples collected pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, and 24 hours post-dose
  Pharmacokinetic analysis by standard model independent methods was performed by a pharmacokineticist using WinNonlin Professional. Actual blood sampling times for ketorolac assay were converted to a time from dosing (elapsed time). Elapsed times were listed by subject for each treatment, together with the individual plasma concentrations of ketorolac.
AUC 0-t (the area under the plasma concentration-time curve (AUC) from time zero to the last quantifiable time point post-dose | All PK parameters were assessed using blood samples collected pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, and 24 hours post-dose
  Pharmacokinetic analysis by standard model independent methods was performed by a pharmacokineticist using WinNonlin Professional. Actual blood sampling times for ketorolac assay were converted to a time from dosing (elapsed time). Elapsed times were listed by subject for each treatment, together with the individual plasma concentrations of ketorolac.
AUCinf (the AUC from time zero to infinity, where possible | All PK parameters were assessed using blood samples collected pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, and 24 hours post-dose
  Pharmacokinetic analysis by standard model independent methods was performed by a pharmacokineticist using WinNonlin Professional. Actual blood sampling times for ketorolac assay were converted to a time from dosing (elapsed time). Elapsed times were listed by subject for each treatment, together with the individual plasma concentrations of ketorolac.
t1/2z (the terminal half-life, where possible | All PK parameters were assessed using blood samples collected pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, and 24 hours post-dose
  Pharmacokinetic analysis by standard model independent methods was performed by a pharmacokineticist using WinNonlin Professional. Actual blood sampling times for ketorolac assay were converted to a time from dosing (elapsed time). Elapsed times were listed by subject for each treatment, together with the individual plasma concentrations of ketorolac.
MRT (the mean residence time) | All PK parameters were assessed using blood samples collected pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, and 24 hours post-dose
  Pharmacokinetic analysis by standard model independent methods was performed by a pharmacokineticist using WinNonlin Professional. Actual blood sampling times for ketorolac assay were converted to a time from dosing (elapsed time). Elapsed times were listed by subject for each treatment, together with the individual plasma concentrations of ketorolac.

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Clarke, BSc MB BS MFPM, Principal Investigator — ICON Development Solutions
Locations (1):
- ICON Development Solutions, Manchester, United Kingdom